CLINICAL TRIAL: NCT04202640
Title: Effectiveness of Mechanical Stimulation on Pain Level and Functional Discomfort Following a Total Mastectomy and Exploratory Axillary Surgery
Brief Title: Mechanical Stimulation on Pain Level and Functional Discomfort After Breast Cancer Surgery
Acronym: PRESSODOU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRESSODOU-1809
Record Dates: First submitted 2019-06-05; First posted 2019-12-17 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Mechanical Stimulation; Mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A - Mechanical Stimulation (Experimental): Patients in this arm will receive, in addition to standard rehabilitation physiotherapy, mechanical stimulation
  Interventions: Procedure: Mechanical Stimulation
- Arm B - Massages (Sham Comparator): Patients in this arm will receive, in addition to standard rehabilitation physiotherapy, massages.
  Interventions: Procedure: Massages

INTERVENTIONS:
Procedure: Mechanical Stimulation — The technique of mechanical stimulation alternates between compression and decompression of the treated area. It aims to reestablish a good blood circulation and lymphatic drainage.
  Arms: Arm A - Mechanical Stimulation
Procedure: Massages — Massages will be carried out according to a specific regime as specified in the study protocol. The massages will be done in 15 sessions of 30 minutes each, done twice a week and will consist of:
  * One part muscle exercise
  * One part skin work (drainage)
  Arms: Arm B - Massages

SUMMARY:
This study evaluates the effectiveness of mechanical stimulation technique compared to massages on pain level and functional discomfort (on the mobility of the shoulder) after 6 months, in breast cancer needing physiotherapy, following a total mastectomy and exploratory axillary surgery.

DETAILED DESCRIPTION:
A prospective, monocentric, randomized, open-labelled in two parallel groups study that evaluates the effectiveness of mechanical stimulation technique compared to massages on pain level and functional discomfort (on the mobility of the shoulder) after 6 months in breast cancer patients needing physiotherapy, following a total mastectomy and exploratory axillary surgery.

Other objectives of the study include:

* Evaluate the efficacy of mechanical stimulation technique compared to massages on pain and functional discomfort (on the mobility of the shoulder) 15 days after the end of physiotherapy.
* Evaluate the impact of mechanical stimulation on the quality of life of patients, in comparison to those receiving massages

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient who had total mastectomy for a breast cancer or pre-cancerous lesions
* Associated with axillary dissection or removal of the sentinel lymph nodes
* Presenting with functional discomfort and/or pain at the control consultation, 3 weeks after the mastectomy and justifying the prescription of physiotherapy
* Possibility to be treated by a physiotherapist who can carry out both techniques and accepts to perform either one of the techniques according to the randomized allocation of the treatment
* Patient covered by the French social security regime
* Signed and informed consent

Exclusion Criteria:

* Immediate breast reconstruction
* Total bilateral mastectomy
* Contraindication to mechanical stimulation technique
* Patient who are planning to move houses in the next 6 months
* Patients under guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Pain level by a numerical scale | 6 months after randomization
  Pain level will be evaluated using a numerical scale of pain
Pain level by using Brief Pain Inventory | 6 months after randomization
  Pain level will be evaluated using Brief Pain Inventory (BPI), there is no global score for this questionnaire, each item must be considered separately.
Pain level by using QDN4 questionnaire | 6 months after randomization
  Pain level will be evaluated using QDN4 questionnaire, which is a pain scale from 0 to 10.
Mobility of the shoulders | 6 months after randomization
  Will be evaluated using the Constant score based on the study by Constant CR, Murley AHG. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res 1987;(214):160-4.
  Pain level, level of daily activities and physical mobility will be assessed with a a scale adapted according to the gender and the patients age.

SECONDARY OUTCOMES:
Pain level by a numerical scale | 15 days after the end of physiotherapy
  Pain level will be evaluated using a numerical scale of pain
Pain level by using Brief Pain Inventory | 15 days after the end of physiotherapy
  Pain level will be evaluated using Brief Pain Inventory (BPI), there is no global score for this questionnaire, each item must be considered separately.
Pain level by using QDN4 questionnaire | 15 days after the end of physiotherapy
  Pain level will be evaluated using QDN4 questionnaire, which is a pain scale from 0 to 10.
Mobility of the shoulders | 15 days after the end of physiotherapy
  Will be evaluated using the Constant score based on the study by Constant CR, Murley AHG. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res 1987;(214):160-4.
  Pain level, level of daily activities and physical mobility will be assessed with a a scale adapted according to the gender and the patients age.
Anxiety | at the baseline and 6 months after
  Will be evaluated using the Hospital Anxiety and Depression Scale (HADS) questionnaire. The questionnaire consists of a list of questions to determine the level of anxiety and depression experienced by the patients. Each question is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression:
  * A score equal to or less than 7 indicates no symptoms,
  * A score of 8 - 10 indicates a questionable symptoms,
  * A score of 11 and above confirms of the presence of anxiety and/or depression symptoms
Quality of Life (QoL) with EORTC-QLQ-C30 | at the baseline and 6 months after
  Will be evaluated using the EORTC-QLQ-C30 questionnaire. This questionnaire aim to assess the quality of life of cancer. It is composed of 30 questions.
  In this questionnaire, the items are scored from 1-4, where 1 = not at all, 2 = a little, 3 = quite a bit and 4 = very much.
  Only 2 items in the EORTC-QLQ-C30 questionnaire are scored from 1-7, where 1 is very poor and 7 is excellent.
Quality of Life (QoL) with EORTC-QLQ-BR23 | at the baseline and 6 months after
  Will be evaluated using the EORTC-QLQ-BR23 questionnaire. This questionnaire aim to assess the quality of life of cancer. It is composed of 23 questions.
  In this questionnaire, the items are scored from 1-4, where 1 = not at all, 2 = a little, 3 = quite a bit and 4 = very much.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia REGIS, MD, Principal Investigator — Centre Oscar Lambret
Locations (2):
- France (2):
  - Centre Oscar Lambret, Lille, Hauts-de-France
  - Centre Hospitalier Universitaire de Lille, Lille

IPD SHARING:
Plan to Share IPD: No